CLINICAL TRIAL: NCT00319696
Title: Long-term Bosentan Open Label Extension of the AC-052-331 Study in Systemic Sclerosis Patients With Ischemic Digital Ulcers
Brief Title: Bosentan in Digital Ulcers
Acronym: RAPIDS 2 OL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-052-333
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Results first posted 2012-08-08 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Digital Ulcers
Keywords: digital ulcers; systemic sclerosis; finger ulcers; bosentan; open label
MeSH Terms: conditions — digital ulcers; Scleroderma, Systemic | interventions — Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bosentan (Experimental): Bosentan 62.5 mg tablets b.i.d. for the first 4 weeks followed by bosentan 125 mg b.i.d. thereafter
  Interventions: Drug: Bosentan 62.5 mg; Drug: Bosentan 125 mg

INTERVENTIONS:
Drug: Bosentan 62.5 mg — Bosentan 62.5-mg oral tablets twice daily (b.i.d.) for 4 weeks (initial dose)
Drug: Bosentan 125 mg — Bosentan 125-mg oral tablets administered b.i.d. (target dose)

SUMMARY:
The aim of the study is to collect long-term efficacy, tolerability and safety data of bosentan in Systemic Sclerosis (SSc) patients suffering from ischemic digital ulcers (DUs).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with SSc according to the classification criteria of the American College of Rheumatology
2. SSc patients with at least one DU at baseline qualifying as a CU (see definition section 3.2.2)
3. CU occurred < 3 months and > 1 week prior to randomization. The subset of patients with SSc felt to be at high risk for DUs will be identified in the screening period but will not be eligible for enrollment until a CU has developed
4. Male or female patients >/= 18 years of age
5. Women of childbearing potential must have a negative pre-treatment pregnancy test and use a reliable method of contraception during study treatment and for at least 3 months after study treatment termination
6. Women not of childbearing potential are defined as postmenopausal (i.e., amenorrhea for at least 1 year), or surgically or naturally sterile
7. Signed informed consent.

Exclusion Criteria:

1. DUs due to condition other than SSc
2. Severe PAH (WHO class III and IV)
3. Systolic blood pressure < 85 mmHg
4. Hemoglobin concentration < 75% of the lower limit of the normal range
5. AST and/or ALT values greater than 3 times the upper limit of normal
6. Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C
7. Severe malabsorption or any severe organ failure (e.g., lung, kidney) or any life-threatening condition
8. Pregnancy or breast-feeding
9. Previous treatment with bosentan
10. Treatment with any of the following: glibenclamide (glyburide), fluconazole, cyclosporine A, tacrolimus and any other calcineurin inhibitor 1 week prior to randomization
11. Local injection of botulinum toxin in an affected finger 1 month prior to randomization
12. Treatment with parenteral prostanoids (prostaglandin E, epoprostenol, treprostinil sodium or other prostacyclin analogs) 3 months prior to randomization
13. Treatment with inhaled or oral prostanoids one month prior to randomization
14. Systemic antibiotics to treat infection of DUs 2 weeks prior to randomization
15. Treatment with phosphodiesterase inhibitors such as sildenafil, except for intermittent treatment of male erectile dysfunction
16. Body weight < 40 kg
17. Patient with conditions that prevent compliance with the protocol or adhering to therapy
18. Patient who received an investigational product within 1 month preceding screening
19. Known hypersensitivity to bosentan or any of the excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2004-07-08 (Actual); Primary Completion 2009-01-22 (Actual); Study Completion 2009-01-22 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 33 centers in 7 countries (Canada, France, Germany, Italy, Switzerland, UK, and USA. The first patient enrolled and started treatment on 8 July 2004 and the last patient enrolled and started treatment on 20 October 2005.
Pre-assignment Details: Patients who completed RAPIDS-2 and who still had digital ulcers (DUs) or developed a new digital ulcer (DU) after the last follow-up visit were eligible. After release of the RAPIDS-2 results, patients who were prematurely discontinued from RAPIDS-2 for treatment failure or, if on placebo, for an adverse event and had DUs were also eligible.
Groups:
- Bosentan: Initial dose: bosentan 62.5 mg twice daily (b.i.d.) for the first 4 weeks. Target dose: bosentan 125 mg b.i.d. thereafter
Period: Overall Study
Arm/Group | Bosentan
Started | 116
Completed | 56
Not Completed | 60
Not completed — Adverse Event | 36
Not completed — withdrawal of consent | 14
Not completed — administrative | 7
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Bosentan
Number analyzed (Participants) | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (12.0)
Age, Customized [Count of Participants; unit: Participants]
  Between 24 and 79 years | 116
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 29
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 11
  France | 10
  Germany | 9
  Italy | 9
  Switzerland | 4
  United Kingdom | 6
  United States | 67
Scleroderma Health Assessment Questionnaire (SHAQ) Individual Domain Score [Mean (Standard Deviation); unit: score on a scale] — SHAQ evaluates physical disability. Patients were instructed to rate their capacity to perform activities of daily living within the previous 7 days by checking one of the following descriptors: "without any difficulty", "with some difficulty," "with much difficulty," or "unable to do," equivalent to scores of 0, 1, 2, and 3, respectively. Items were categorized into 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities.
  score on a scale
    Dressing | 1.3 (0.9)
    Arising | 0.5 (0.8)
    Eating | 1.5 (1.0)
    Walking | 0.5 (0.7)
    Hygiene | 0.9 (1.0)
    Reach | 1.1 (0.9)
    Grip | 1.1 (0.8)
    Activity | 1.0 (0.9)
Overall hand pain [Mean (Standard Deviation); unit: mm] — Overall hand pain related to finger ulcers was assessed by the patient using a Visual Analogue Scale. Patients were instructed to score their pain by marking on the continuous 10-cm scale, where 0 (left) was no pain and 100 (right) very severe pain, in response to the question, "How much pain have you had because of your finger ulcers in the past week?" The investigator measured the distance in millimeters between 0 and the patient mark with the ruler provided and recorded the distance.
  mm | 58.62 (29.80)
United Kingdom Scleroderma Functional Score (UKFS) [Mean (Standard Deviation); unit: score on a scale] — UKFS relates to upper and lower extremity function and muscle weakness. For each item, the patient indicated the responses that best described their current ability: "able to perform in a normal manner," "able to perform with alteration in style," "can only manage with difficulty," and "impossible to achieve." Each response was given an integer from 0 (able to perform in a normal manner) to 3 (impossible to achieve), and the sum of individual responses provided an overall score of 0 to 33. Missing values were replaced with the worst value the patient reported on the other items at that visit.
  score on a scale | 11.06 (7.50)

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete Healing of Each Baseline DU
Time Frame: Baseline to healing
Population: Complete healing of each baseline was not calculated due to the lack of effect on healing variables seen in the previous placebo-controlled study (RAPIDS 2). In consequence, the endpoint on time to complete healing of baseline DUs was not evaluated.
Arm/Group | Bosentan
Number analyzed (Participants) | 0

2. Primary Outcome: Time to Complete Healing of Each New DU
Time Frame: New DU occurence to healing
Population: Complete healing of each new DU was not calculated due to the lack of effect on healing variables seen in the previous placebo-controlled study (RAPIDS 2). In consequence, the endpoint on DU healing originally planned time to complete healing of new DUs was not evaluated.
Arm/Group | Bosentan
Number analyzed (Participants) | 0

3. Primary Outcome: Mean Change From Baseline at Each 16 Week Interval up to Week 80 in Scleroderma Health Assessment Questionnaire (SHAQ) Individual Domain Score: Dressing
Description: SHAQ evaluates physical disability. Patients were instructed to rate their capacity to perform activities of daily living within the previous 7 days by checking one of the following descriptors: "without any difficulty", "with some difficulty," "with much difficulty," or "unable to do," equivalent to scores of 0, 1, 2, and 3, respectively. Items were categorized into 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities.
Time Frame: 80 weeks
Population: number of participants at baseline, week 16, week 32, week 48, week 64, and week 80 was 116, 99, 93, 85, 82, and 78, respectively
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Bosentan
Number analyzed (Participants) | 116
scores on a scale
  change from baseline to week 16 | -0.3 (0.6)
  change from baseline to week 32 | -0.2 (0.7)
  change from baseline to week 48 | -0.1 (0.7)
  change from baseline to week 64 | -0.1 (0.7)
  change from baseline to week 80 | -0.1 (0.7)

4. Primary Outcome: Mean Change From Baseline at Each 16 Week Interval up to Week 80 in Scleroderma Health Assessment Questionnaire (SHAQ) Individual Domain Score: Arising
Description: as for outcome 3
Time Frame: 80 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Bosentan
Number analyzed (Participants) | 116
scores on a scale
  change from baseline to week 16 | 0.0 (0.6)
  change from baseline to week 32 | -0.0 (0.6)
  change from baseline to week 48 | 0.1 (0.6)
  change from baseline to week 64 | 0.1 (0.7)
  change from baseline to week 80 | 0.1 (0.6)

5. Primary Outcome: Mean Change From Baseline at Each 16 Week Interval up to Week 80 in Scleroderma Health Assessment Questionnaire (SHAQ) Individual Domain Score: Eating
Description: as for outcome 3
Time Frame: 80 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Bosentan
Number analyzed (Participants) | 116
scores on a scale
  change from baseline to week 16 | -0.2 (0.6)
  change from baseline to week 32 | -0.1 (0.7)
  change from baseline to week 48 | -0.2 (0.7)
  change from baseline to week 64 | -0.1 (0.6)
  change from baseline to week 80 | -0.1 (0.7)

6. Primary Outcome: Mean Change From Baseline at Each 16 Week Interval up to Week 80 in Scleroderma Health Assessment Questionnaire (SHAQ) Individual Domain Score: Walking
Description: as for outcome 3
Time Frame: 80 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Bosentan
Number analyzed (Participants) | 116
scores on a scale
  change from baseline to week 16 | -0.1 (0.6)
  change from baseline to week 32 | 0.0 (0.7)
  change from baseline to week 48 | 0.1 (0.7)
  change from baseline to week 64 | 0.1 (0.8)
  change from baseline to week 80 | 0.1 (0.8)

7. Primary Outcome: Mean Change From Baseline at Each 16 Week Interval up to Week 80 in Scleroderma Health Assessment Questionnaire (SHAQ) Individual Domain Score: Hygiene
Description: as for outcome 3
Time Frame: 80 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Bosentan
Number analyzed (Participants) | 116
scores on a scale
  change from baseline to week 16 | -0.0 (0.7)
  change from baseline to week 32 | -0.0 (0.8)
  change from baseline to week 48 | -0.0 (0.8)
  change from baseline to week 64 | 0.1 (0.7)
  change from baseline to week 80 | 0.2 (0.8)

8. Primary Outcome: Mean Change From Baseline at Each 16 Week Interval up to Week 80 in Scleroderma Health Assessment Questionnaire (SHAQ) Individual Domain Score: Reach
Description: as for outcome 3
Time Frame: 80 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Bosentan
Number analyzed (Participants) | 116
scores on a scale
  change from baseline to week 16 | -0.1 (0.7)
  change from baseline to week 32 | 0.0 (0.7)
  change from baseline to week 48 | 0.0 (0.8)
  change from baseline to week 64 | 0.1 (0.8)
  change from baseline to week 80 | 0.0 (0.7)

9. Primary Outcome: Mean Change From Baseline at Each 16 Week Interval up to Week 80 in Scleroderma Health Assessment Questionnaire (SHAQ) Individual Domain Score: Grip
Description: as for outcome 3
Time Frame: 80 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Bosentan
Number analyzed (Participants) | 116
scores on a scale
  change from baseline to week 16 | -0.1 (0.7)
  change from baseline to week 32 | -0.2 (0.7)
  change from baseline to week 48 | -0.1 (0.7)
  change from baseline to week 64 | -0.1 (0.7)
  change from baseline to week 80 | -0.1 (0.7)

10. Primary Outcome: Mean Change From Baseline at Each 16 Week Interval up to Week 80 in Scleroderma Health Assessment Questionnaire (SHAQ) Individual Domain Score: Activity
Description: as for outcome 3
Time Frame: 80 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Bosentan
Number analyzed (Participants) | 116
scores on a scale
  change from baseline to week 16 | -0.2 (0.5)
  change from baseline to week 32 | -0.1 (0.7)
  change from baseline to week 48 | -0.1 (0.7)
  change from baseline to week 64 | -0.1 (0.7)
  change from baseline to week 80 | -0.1 (0.6)

11. Primary Outcome: Mean Changes From Baseline at Each 16 Week Interval up to Week 80 in Overall Hand Pain Related to Finger Ulcers
Description: Overall hand pain related to finger ulcers was assessed by the patient using a Visual Analogue Scale. Patients were instructed to score their pain by marking on the continuous 10-cm scale, where 0 (left) was no pain and 100 (right) very severe pain, in response to the question, "How much pain have you had because of your finger ulcers in the past week?" The investigator measured the distance in millimeters between 0 and the patient mark with the ruler provided and recorded the distance.
Time Frame: 80 weeks
Population: number of participants at baseline, week 16, week 32, week 48, week 64, and week 80 was 110, 94, 89, 81, 76, and 73, respectively
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bosentan
Number analyzed (Participants) | 116
mm
  change from baseline to week 16 | -21.59 (28.02)
  change from baseline to week 32 | -28.16 (32.64)
  change from baseline to week 48 | -21.90 (32.09)
  change from baseline to week 64 | -22.96 (33.27)
  change from baseline to week 80 | -24.29 (36.55)

12. Primary Outcome: Mean Change From Baseline at Each 16 Week Interval up to Week 80 in the UK Systemic Sclerosis Functional Score (UKFS)
Description: UKFS relates to upper and lower extremity function and muscle weakness. For each item, the patient indicated the responses that best described their current ability: "able to perform in a normal manner," "able to perform with alteration in style," "can only manage with difficulty," and "impossible to achieve." Each response was given an integer from 0 (able to perform in a normal manner) to 3 (impossible to achieve), and the sum of individual responses provided an overall score of 0 to 33. Missing values were replaced with the worst value the patient reported on the other items at that visit.
Time Frame: 80 weeks
Population: number of participants at baseline, week 16, week 32, week 48, week 64, and week 80 was 116, 98, 93, 84, 82, and 78, respectively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bosentan
Number analyzed (Participants) | 116
score on a scale
  change from baseline to week 16 | -1.37 (3.64)
  change from baseline to week 32 | -1.25 (4.01)
  change from baseline to week 48 | -0.89 (4.98)
  change from baseline to week 64 | -1.17 (4.00)
  change from baseline to week 80 | -0.45 (4.66)

13. Primary Outcome: Total Number of New Digital Ulcers (DUs) Per Patient Observed by the Investigator at Planned Visits
Description: The total number of new DUs per patient observed by the investigator at planned visits and new transient DUs recorded in the patient diary (a patient diary was used to record DUs that might appear and disappear between two planned visits) were assessed at each clinic visit
Time Frame: At planned visits up to week 80
Population: One patient did not have a DU at baseline (number of patients assessed at Weeks 0-4,4-8,8-16,16-24,24-32,32-40,40-48,48-56,56-64,64-72, and 72-80 were 114, 107, 103, 100, 97, 94, 88, 87, 86, 86, and 83, respectively.
Measure: Number; unit: number of new digital ulcers
Groups:
- 0 New Ulcers; At Least 1 New Ulcer; At Least 2 New Ulcers; At Least 3 New Ulcers; At Least 4 New Ulcers; At Least 5 New Ulcers: Number of new DUs includes the new number at each visit and the transient ulcers between visits.
Arm/Group | 0 New Ulcers | At Least 1 New Ulcer | At Least 2 New Ulcers | At Least 3 New Ulcers | At Least 4 New Ulcers | At Least 5 New Ulcers
Number analyzed (Participants) | 115 | 115 | 115 | 115 | 115 | 115
number of new digital ulcers
  Week 0-4 | 85 | 29 | 17 | 6 | 4 | 3
  Week 4-8 | 73 | 34 | 15 | 6 | 4 | 3
  Week 8-16 | 63 | 40 | 22 | 9 | 7 | 5
  Week 16-24 | 64 | 36 | 17 | 11 | 4 | 2
  Week 24-32 | 56 | 41 | 22 | 12 | 8 | 4
  Week 32-40 | 59 | 35 | 15 | 7 | 5 | 4
  Week 40-48 | 52 | 36 | 20 | 11 | 5 | 3
  Week 48-56 | 50 | 37 | 18 | 13 | 7 | 5
  Week 56-64 | 48 | 38 | 14 | 7 | 4 | 3
  Week 64-72 | 51 | 35 | 24 | 15 | 10 | 8
  Week 72-80 | 51 | 32 | 18 | 9 | 4 | 2

14. Secondary Outcome: Adverse Events up to 24 Hours After Last Study Medication
Description: Number of patients with at least one treatment-emergent adverse event. All adverse events that occurred after study drug initiation and up to 24 hours after study drug discontinuation were to be recorded.
Time Frame: 80 weeks
Population: Study population
Measure: Number; unit: participants
Arm/Group | Bosentan
Number analyzed (Participants) | 116
participants | 111

15. Secondary Outcome: Adverse Events Leading to Permanent Discontinuation of the Study Medication
Description: Number of patients with an adverse event leading to permanent discontinuation of the study treatment
Time Frame: 80 weeks
Population: Study population
Measure: Number; unit: participants
Arm/Group | Bosentan
Number analyzed (Participants) | 116
participants | 36

16. Secondary Outcome: Serious Adverse Events up to 28 Days After Last Study Medication
Description: Number of patients with at least one treatment-emergent serious adverse event (TESAE) were reported. TESAEs are serious AEs that occurred after study drug initiation and up to 28 days after study drug discontinuation. More details on the SAEs are provided in the specific Adverse Events Section
Time Frame: 80 weeks
Measure: Number; unit: Participants
Arm/Group | Bosentan
Number analyzed (Participants) | 116
Participants | 45

ADVERSE EVENTS:
Time Frame: 80 weeks
Description: Treatment-emergent adverse events
Arm/Group | Bosentan
All-Cause Mortality (participants affected / at risk) | 6/116
Serious Adverse Events (participants affected / at risk) | 45/116
Other Adverse Events (participants affected / at risk) | 111/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosentan (N=116)
PNEUMONIA (Infections and infestations) | 6
INFECTED SKIN ULCER (Infections and infestations) | 4
CELLULITIS (Infections and infestations) | 2
DEVICE RELATED INFECTION (Infections and infestations) | 2
SEPSIS (Infections and infestations) | 2
ABSCESS LIMB (Infections and infestations) | 1
APPENDICITIS (Infections and infestations) | 1
BRONCHITIS (Infections and infestations) | 1
CATHETER SITE INFECTION (Infections and infestations) | 1
DIVERTICULITIS (Infections and infestations) | 1
GANGRENE (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 1
HEPATITIS B (Infections and infestations) | 1
HERPES ZOSTER (Infections and infestations) | 1
INFLUENZA (Infections and infestations) | 1
LOBAR PNEUMONIA (Infections and infestations) | 1
LOCALISED INFECTION (Infections and infestations) | 1
OSTEOMYELITIS (Infections and infestations) | 1
VIRAL PERICARDITIS (Infections and infestations) | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 2
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 2
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 1
FAECALOMA (Gastrointestinal disorders) | 1
GASTRITIS (Gastrointestinal disorders) | 1
GASTROINTESTINAL MOTILITY DISORDER (Gastrointestinal disorders) | 1
ILEUS (Gastrointestinal disorders) | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 1
OESOPHAGITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2
SCLERODERMA (Musculoskeletal and connective tissue disorders) | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1
MYOSITIS (Musculoskeletal and connective tissue disorders) | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1
SYSTEMIC SCLEROSIS (Musculoskeletal and connective tissue disorders) | 1
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 1
ADVERSE DRUG REACTION (General disorders) | 2
CHEST PAIN (General disorders) | 2
DEVICE DISLOCATION (General disorders) | 1
DRUG WITHDRAWAL SYNDROME (General disorders) | 1
IMPAIRED HEALING (General disorders) | 1
PAIN (General disorders) | 1
SUPRAPUBIC PAIN (General disorders) | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 5
PYODERMA GANGRENOSUM (Skin and subcutaneous tissue disorders) | 1
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1
SKIN NECROSIS (Skin and subcutaneous tissue disorders) | 1
PERIPHERAL ISCHAEMIA (Vascular disorders) | 4
EXTREMITY NECROSIS (Vascular disorders) | 1
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 1
HYPOTENSION (Vascular disorders) | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1
CARDIAC ARREST (Cardiac disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1
MYOCARDITIS (Cardiac disorders) | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1
DIZZINESS POSTURAL (Nervous system disorders) | 1
HYPOAESTHESIA (Nervous system disorders) | 1
LUMBAR RADICULOPATHY (Nervous system disorders) | 1
PARAESTHESIA (Nervous system disorders) | 1
ARTHRODESIS (Surgical and medical procedures) | 1
FINGER AMPUTATION (Surgical and medical procedures) | 1
FOOT AMPUTATION (Surgical and medical procedures) | 1
HIP ARTHROPLASTY (Surgical and medical procedures) | 1
LUNG TRANSPLANT (Surgical and medical procedures) | 1
REVISION OF INTERNAL FIXATION (Surgical and medical procedures) | 1
ASBESTOSIS (Injury, poisoning and procedural complications) | 1
JOINT INJURY (Injury, poisoning and procedural complications) | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 1
ANAEMIA (Blood and lymphatic system disorders) | 2
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1
SCLERODERMA RENAL CRISIS (Renal and urinary disorders) | 2
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1
MALNUTRITION (Metabolism and nutrition disorders) | 1
ALCOHOLIC PSYCHOSIS (Psychiatric disorders) | 1
DEPRESSION (Psychiatric disorders) | 1
HEPATIC ENZYME INCREASED (Investigations) | 1
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bosentan (N=116)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 26
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 24
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 22
DIARRHOEA (Gastrointestinal disorders) | 21
INFECTED SKIN ULCER (Infections and infestations) | 21
LOCALISED INFECTION (Infections and infestations) | 17
COUGH (Respiratory, thoracic and mediastinal disorders) | 15
HEADACHE (Nervous system disorders) | 14
RASH (Skin and subcutaneous tissue disorders) | 14
NASOPHARYNGITIS (Infections and infestations) | 13
NAUSEA (Gastrointestinal disorders) | 13
OEDEMA PERIPHERAL (General disorders) | 13
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 13
PRURITUS (Skin and subcutaneous tissue disorders) | 13
LIVER FUNCTION TEST ABNORMAL (Investigations) | 12
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 11
ANAEMIA (Blood and lymphatic system disorders) | 11
DYSPHAGIA (Gastrointestinal disorders) | 11
FATIGUE (General disorders) | 11
BRONCHITIS (Infections and infestations) | 10
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 10
INSOMNIA (Psychiatric disorders) | 10
SINUSITIS (Infections and infestations) | 10
INFLUENZA (Infections and infestations) | 9
PYREXIA (General disorders) | 9
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 8
TENDONITIS (Musculoskeletal and connective tissue disorders) | 8
URINARY TRACT INFECTION (Infections and infestations) | 8
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 7
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7
CELLULITIS (Infections and infestations) | 7
GASTROENTERITIS VIRAL (Infections and infestations) | 7
ASTHENIA (General disorders) | 6
DIZZINESS (Nervous system disorders) | 6
HAEMOGLOBIN DECREASED (Investigations) | 6
HERPES ZOSTER (Infections and infestations) | 6
MOUTH ULCERATION (Gastrointestinal disorders) | 6
WEIGHT DECREASED (Investigations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related article or abstract written independently by investigators should be submitted to Actelion for review at least 60 days prior to submission for publication or presentation.